CLINICAL TRIAL: NCT06101914
Title: Evaluating the Occurrence of Engagement Patterns and Participation Trends Among Patients in Treatment Resistant Depression
Brief Title: Studying Patterns in Patient Engagement Among Treatment Resistant Depression Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Power Life Sciences Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 64175778
Record Dates: First submitted 2023-10-20; First posted 2023-10-26 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Treatment Resistant Depression
Keywords: treatment resistant depression
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Clinical studies, with a distinct focus on treatment resistant depression, play a crucial role in evaluating the safety and effectiveness of novel treatments. These trials serve as instrumental means to determine whether new medications surpass conventional therapies, providing substantial evidence for their broader adoption.

The primary objective is to meticulously scrutinize trial completion rates and voluntary withdrawals within this specific patient group.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of treatment resistant depression
* Aged ≥ 18 years old and ability to provide written informed consent obtained prior to participation in the study and any related procedures being performed
* No prior treatment for treatment resistant depression

Exclusion Criteria:

* Enrolled in another research study
* Inability to provide written informed consent
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Treatment resistant depression patients who are actively considering enrolling in a clinical trial for the said condition, but have not yet completed enrollment and randomization phases.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Rate of patients who decide to enroll in a treatment resistant depression clinical research. | 3 months
Number of treatment resistant depression study participants who remain in clinical study until completion. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Gill, Study Director — Power Life Sciences Inc.
Locations (1):
- Power Life Sciences, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lundberg J, Cars T, Loov SA, Soderling J, Sundstrom J, Tiihonen J, Leval A, Gannedahl A, Bjorkholm C, Sjalin M, Hellner C. Association of Treatment-Resistant Depression With Patient Outcomes and Health Care Resource Utilization in a Population-Wide Study. JAMA Psychiatry. 2023 Feb 1;80(2):167-175. doi: 10.1001/jamapsychiatry.2022.3860. PMID 36515938
- [Background] Perez-Sola V, Roca M, Alonso J, Gabilondo A, Hernando T, Sicras-Mainar A, Sicras-Navarro A, Herrera B, Vieta E. Economic impact of treatment-resistant depression: A retrospective observational study. J Affect Disord. 2021 Dec 1;295:578-586. doi: 10.1016/j.jad.2021.08.036. Epub 2021 Aug 27. PMID 34509073
- [Background] Wilkowska A, Wlodarczyk A, Galuszko-Wegielnik M, Wiglusz MS, Cubala WJ. Intravenous Ketamine Infusions in Treatment-Resistant Bipolar Depression: An Open-Label Naturalistic Observational Study. Neuropsychiatr Dis Treat. 2021 Aug 14;17:2637-2646. doi: 10.2147/NDT.S325000. eCollection 2021. PMID 34421299

DOCUMENTS (1):
  • Informed Consent Form (2023-10-20): https://cdn.clinicaltrials.gov/large-docs/14/NCT06101914/ICF_000.pdf